CLINICAL TRIAL: NCT01269229
Title: A Phase 2 Trial of Neoadjuvant FOLFOX6 With Short Course Radiotherapy in Patients With Unresectable Rectal Cancer and Liver Metastasis
Brief Title: A Trial of Neoadjuvant FOLFOX6 With Short Course Radiotherapy in Patients With Unresectable Rectal Cancer and Liver Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0522
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: folfox — FOLFOX: Day1- Oxaliplatin 85mg/m2, Leucovorin 200mg/m2, 5-FU 400mg/m2 IV bolus -> 2400mg/m2 46hrs continuous
Radiation: short course Radiotherapy — After FOLFOX 4cycle, subject have short course RTx 5Gy at once this should be continuing for 5days so that subject should have 25Gy within 5days. Then, subjects have another 4 cycle of FOLFOX and evaluate cancer for resection.

SUMMARY:
The purpose of this study is the increase of resection rate of primary cancer in rectal after short course radiotherapy without interrupt chemotherapy schedule during the period of chemotherapy. The subject should have the pathologically confirmed for unresectable (impossible to try Total mesorectal excision) rectal cancer with liver metastasis.

This trial contributes to save the time for decreasing primary tumor in rectal and metastasis cancer to whole body after short course radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject whom should have the pathologically confirmed for unresectable (impossible to try Total mesorectal excision) rectal cancer with liver metastasis.
* Over 18 years
* ECOG 0-1
* Proper organ function (hepatic transaminases : < ULN ⅹ5, Bilirubin: < ULNⅹ2, creatinine (serum): < ULNⅹ 1.5, PLT > 100,000Ul, ANC > 1,500/Ul
* more than one target lesion (standard by RECIST 1.0)
* Who should sign on the Informed consent form before participate the trial.

Exclusion Criteria:

* Metastasis in other organ except liver (No matter whether have resection or not)
* Chronic active hepatitis or cirrhosis
* History of treatment for colorectal cancer
* Subject pregnant or breast feeding
* Uncontrolled disease (eg. infection, hypertension, heart failure, Myocardial Infarction within 6months)
* Have been used FOLFOX as an adjuvant therapy
* Have had adjuvant therapy within 6months
* Uncontrolled peripheral nerve infection
* Alcoholic or drug addict
* Subject currently is enrolled in or ≤30 days from ending other clinical trial.
* History of other type of cancer except resolved from skin cancer and cervical cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
complete resection (R0) rate for rectal and liver lesions. | after surgical resection
  Complete resection (R0 resection) is defined as no residual cancer cells in the resection margn both primary recal mass and liver metastases after simultaneous surgical resection.

SECONDARY OUTCOMES:
Response rate (RECIST V1.0) | every 4 cycles
Overall survival rate | participants will be followed until death
Progression free survival time | participants will be followed until disease progression or death
Toxicity profile | participants will be followed until disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea